CLINICAL TRIAL: NCT05956054
Title: A Comparison of Intravascular Penetration With Curved Needle and Straight Needle During Sacral 1 Transforaminal Epidural Block
Brief Title: A Comparison of Intravascular Penetration With Curved Needle and Straight Needle During S1 STE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Kyungpook National University Chilgok Hospital (Other)
Responsible Party: Principal Investigator, Jinyoung Oh, assistant professor, Kyungpook National University Chilgok Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: 2023-04-018-001
Record Dates: First submitted 2023-07-13; First posted 2023-07-21 (Actual); Last update posted 2023-07-21 (Actual); Status verified 2023-07

CONDITIONS: S1 Transforaminal Epidural Injection
Keywords: S1 transforaminal epidural injection; curved needle

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- S1 transforaminal injection with a straight needle (Active Comparator)
  Interventions: Other: needle type
- S1 transforaminal injection with a curved needle (Experimental)
  Interventions: Other: needle type

INTERVENTIONS:
Other: needle type — straight or curved

SUMMARY:
The goal of this observational study is to compare in intravasation rate during S1 transforaminal epidural injection between using a straight needle and a curved needle. The main question it aims to answer are:

The main question it aims to answer is:

• whether there is a difference in intravascular rate between using a straight needle and a curved needle in S1 transforaminal epidural injection

Participants in this study will be randomly assigned to receive an S1 transforaminal epidural injection using either a straight needle or a curved needle. The researchers will then observe the intravasation rate and compare it between the two groups.

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled for a lumbar 1 epidural nerve block in the outpatient department of anesthesiology and pain medicine at Kyungpook National University Hospital.

Exclusion Criteria:

1. Patients with a history of allergy to local anesthetics or steroids
2. Patients with a history of allergy to contrast media
3. Patients with a bleeding tendency
4. Patients with symptoms of infection in the sacroiliac region
5. Patients under 18 years of age or over 80 years of age
6. Patients who are pregnant or planning to become pregnant
7. Other medically incapable of consent, such as the mentally retarded.

Translated with www.DeepL.com/Translator (free version)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Estimated)
Dates: Start 2023-06-22 (Actual); Primary Completion 2024-04-02 (Estimated); Study Completion 2024-04-02 (Estimated)

PRIMARY OUTCOMES:
Intravasation rate | in the procedure

CONTACTS AND LOCATIONS:
Locations (1):
- Kyungpook National University Hospital, Daegu, South Korea